CLINICAL TRIAL: NCT02762318
Title: Identification and Characterization of Bone-related Genetic Variants in Families
Status: Terminated | Type: Observational
Why Stopped: Lack of funding
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-00098
Record Dates: First submitted 2015-12-16; First posted 2016-05-04 (Estimated); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Skeletal Dysplasia
MeSH Terms: conditions — Mucopolysaccharidosis IV | interventions — DNA

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Cheek swab (optional)
  [If for any reason, the blood sample cannot be obtained, a swab will be applied to the inside of the cheek to obtain saliva]
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Samples With DNA — After consenting, all subjects have to undergo the following procedures:
  Up to 25 ml of blood will be withdrawn. If for any reason, the blood sample cannot be obtained, a swab will be applied to the inside of the cheek to obtain saliva.
  A questionnaire will be used to collect information about individual A routine physical exam will be performed. The subject's medical record will be reviewed To well document some of the specific phenotypes and conditions, physicians might take photographs of the affected body area.
  For secondary subjects (relatives or family members), normal examination and routine lab tests/ imagining will be done if needed as per the related standard care.

SUMMARY:
Identify novel genetic variants causing skeletal dysplasia in Qatari populations and to additionally develop an understanding of how those variants influence skeletal biology at a molecular and cellular level.

DETAILED DESCRIPTION:
To identify novel genetic variants causing skeletal dysplasia in Qatari populations and to additionally develop an understanding of how those variants influence skeletal biology at a molecular and cellular level.

Achieving this goal will be split into two aims:

* Aim 1: Perform a clinical characterization of a study group of patients with various forms of skeletal dysplasia seen in pediatric orthopedics clinic at Hamad Medical center, HMC. This will be followed by whole exome or genome sequencing and analysis to search for novel pathogenic variants responsible for the clinical presentation of these patients
* Aim 2: The genes and variants identified in Aim 1 will be characterized to determine their effects on osteoblast and chondrocyte differentiation and function.

All the subjects will be recruited from the pool of patients seen by the Pediatric Orthopedic Consultants at the Bone and Joint Institute. Subjects will be coming to the clinic for their standard care. They will be identified during that visit as candidates for the study. They will then be told about the study by their physicians. If a patient is interested in participation, the physician will introduce the CRC to him/her who will proceed with the consent process.

Consenting and the study procedures might be performed during that same visit if time allows, or in a new scheduled visit arranged at that time.

This research will also involve a pedigree creation. Secondary subjects (family members or relatives) will be told about the study by the research subject. The secondary subject will be able to read a copy of the consent form, think of his participation, and if interested they will be told to contact the Investigators. A suitable time will then be arranged, by an appropriate member of the research team, for the secondary subject to visit the clinic in order to proceed with the consent process and the study procedures.

ELIGIBILITY:
Inclusion Criteria:

1. All included individuals must provide informed consent
2. Patients identified to have a skeletal dysplasia
3. All ethnic backgrounds are acceptable
4. Disease must be genetic with no evident environmental cause.
5. Evidence of Mendelian Transmission determined by fulfilling one of the following criteria:

   1. Multiple affected family members (at least first-degree relative with disease)
   2. History of consanguinity
   3. Severe disease in newborn in the absence of family history
   4. Syndromic disease in single individuals
   5. Congenital abnormality affecting major organ system(s)
   6. Mendelianized extremes of common disease (e.g. bilateral developmental dysplasia of the hip)
6. All ages will be included
7. Rare diseases or rare forms of known diseases
8. Unaffected family members or relatives of the individual with the primary syndrome

Exclusion Criteria:

1. Individuals who do not consent will not be included
2. Individuals for which a molecular diagnosis has already been established by alternative method (e.g. karyotype or known gene mutation)
3. Diseases for which an environmental factor is most likely the cause (e.g. Traumatic bone injury or Rickets)
4. Diseases of which late age of onset rule out Mendelian transmission
5. Common Diseases for which late age of onset rule out Mendelian transmission (e.g.Osteoporosis)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All our subjects will be recruited from the pool of patients seen by the Pediatric Orthopedic Consultants at the Bone and Joint Institute. Subjects will be coming to the clinic for their standard care. They will be identified during that visit as candidates for the study.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-12; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Clinical assessement of a study group of patients with various forms of skeletal dysplasia, followed by identification of novel pathogenic variants using whole exome/genome sequencing. | 2-3 years
  Patients will be selected for the study and will undergo:
  Phenotyping by a combination of clinical history taking and examination, determination of bone mass, laboratory studies, Full exome sequencing Lastly, the variants present in each exome will be determined, and these variants will be classified according to their likelihood of being pathogenic.

SECONDARY OUTCOMES:
Biochemical and cellular characterization of the putative causative genes. | 1-2 year
  Chondrocytes or osteoblasts will be used to measure the following:
  Putative gene expression in the skeletal system, How they influence osteoblast and chondrocyte differentiation how they alter the activity of the key molecular pathways governing the activity of osteoblasts and chondrocytes,

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Yes
To facilitate future genetic diagnostics related to skeletal dysplasias, the variants identified and their classifications will be shared in Gulf-based health forums and the international online databases of clinically significant genetic variation in humans (ie Clinvar, dbSNP). The data gathered regarding the spectrum of disorders identified will be similarly disseminated. HMC-affiliated investigators will use the data generated for poster and oral presentations at international meetings. Similarly, the genetic data will be likewise shared at the relevant local and international meetings. Most importantly, we are committed to publishing the results in a timely fashion in the biomedical literature, aiming for publications in high quality, high impact, peer reviewed journals. All original data and reagents generated will be made available to other investigators according to the conventions of biomedical science.